CLINICAL TRIAL: NCT04394754
Title: Assessing the Efficacy of Digital Health Technology in the Management of Congestive Heart Failure: An Evaluation of Three Novel Digital Health Products
Brief Title: Evaluating Efficacy of Digital Health Technology in the Treatment of Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boehringer Ingelheim (Industry); ZS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000027325
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Congestive Heart Failure
Keywords: Digital Health
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Control (No Intervention): Patients will receive usual care and no digital health device.
- BodyPort (Experimental): Patients will receive the BodyPort device.
  Interventions: Device: BodyPort
- Noom (Experimental): Patients will receive a subscription to the Noom platform.
  Interventions: Other: Noom
- Conversa (Experimental): Patients will receive a subscription to the Conversa platform.
  Interventions: Other: Conversa

INTERVENTIONS:
Device: BodyPort — Patients will receive BodyPort, a smart scale that provides advanced cardiac monitoring.
  Arms: BodyPort
Other: Noom — Patients will receive a subscription to use Noom, a personalized diet and weight management application.
  Arms: Noom
Other: Conversa — patients will receive a subscription to use Conversa, a personalized automated coaching and motivational application.
  Arms: Conversa

SUMMARY:
The purpose of this study is to determine the efficacy of three novel digital health technologies versus usual care in the management of congestive heart failure, as assessed by a primary outcome of improvement in quality of life, and a variety of secondary outcomes that include metrics measuring patient and provider satisfaction, clinical efficiency, and patient outcomes.

DETAILED DESCRIPTION:
Heart failure is the most common cause of mortality and morbidity in the United States and in Western Europe. However, patient etiology and prognosis varies considerably, and guidance about how to best treat patients has relied on large clinical trials that only include snapshots of the syndrome (at the time the patient interaction with the healthcare system). It remains to be seen whether behavioral interventions can improve patient engagement, increase self-management of the conditions, and thus improve overall clinical outcomes.

Digital health technologies have a great potential to streamline and optimize the clinical management of heart failure. Such technologies can take the form of mobile applications or wearable devices that may provide both patients and providers with valuable real-time information about patient status and cardiovascular health, provide automated patient-tailored coaching and motivational tools, or a mix of both. Integration of these technologies into healthcare systems may allow for genuine engagement of the patient in their own care and management of their disease and/or enhance clinical decision making. To date, no prior study has comprehensively examined the ability of digital heath technologies to improve self-management of heart failure or subsequent clinical outcomes.

This study is an unblinded, 4-arm, parallel group randomized controlled trial to measure the efficacy of four digital health technologies in improving the management of care and quality of life of patients with congestive heart failure (CHF). Patients actively managed by one of Yale New Haven Hospital's heart failure-based clinics will be eligible for this study and approached for consent. Enrolled subjects will be randomized to one of four groups: a control (usual care) arm, or to one of three intervention arms, each of which assesses one of three digital health technologies. These technologies are:

* BodyPort: A data-driven smart scale that provides enhanced cardiac monitoring and risk assessment data.
* Noom: A live, data-driven coaching application providing personalized diet and weight management.
* Conversa: An automated conversational platform providing patient motivation and educational tools for CHF management.

Patients will be enrolled in the study for 6 months. The first three months will typically involve active clinic management and will be the point of our primary outcome assessment, while the final three months will assess stability of effect on patient care and outcomes.

The primary outcome is the rate of improvement in quality of life after 90 days post-enrollment, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ). A variety of prespecified secondary outcomes will be measured to determine effects on patient outcomes, quality of care, clinical efficiency, and provider and patient satisfaction with the product.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 and less than 80 years of age
* Enrolled in one of Yale New Haven Hospital's Disease Management or Heart Failure-focused cardiology clinics
* Diagnosed with congestive heart failure (preserved or reduced ejection fraction with or without diabetes)

Exclusion Criteria:

* Class IV heart failure
* Stage 4 or end stage renal disease (eGFR < 30)
* Recipient of a heart transplant of ventricular assist device
* Under hospice care
* Dementia
* Incarceration
* Pregnancy
* Currently homeless or residing in an unstable living situation (i.e., transitional housing, rehab facility, etc.)
* Inability to consent
* Currently enrolled in a study investigating a digital health product or technology
* Life expectancy of less than 6 months as determined by clinical judgement of primary treating physician
* weight greater than 400 pounds
* unable to stand straight up for 30 seconds without assistance, such as from a cane, walker, or wall.
* non-English speaking

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Wilson, MD MSCE, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data underlying results will be made available upon publication in an appropriate database.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication; indefinitely

REFERENCES:
- [Derived] Victoria-Castro AM, Martin ML, Yamamoto Y, Melchinger H, Weinstein J, Nguyen A, Lee KA, Gerber B, Calderon F, Subair L, Lee V, Williams A, Shaw M, Arora T, Garcez A, Desai NR, Ahmad T, Wilson FP. Impact of Digital Health Technology on Quality of Life in Patients With Heart Failure. JACC Heart Fail. 2024 Feb;12(2):336-348. doi: 10.1016/j.jchf.2023.09.022. Epub 2023 Nov 8. PMID 37943227

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | BodyPort | Noom | Conversa
Started | 44 | 46 | 46 | 46
Completed | 36 | 39 | 38 | 38
Not Completed | 8 | 7 | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | BodyPort | Noom | Conversa | Total
Number analyzed (Participants) | 44 | 46 | 46 | 46 | 182
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [50 to 65.5] | 59 [54 to 66] | 62 [54 to 70] | 62.5 [55 to 72] | 61 [53 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 21 | 16 | 69
  Male | 31 | 27 | 25 | 30 | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-hispanic white | 24 | 30 | 27 | 25 | 106
  Non-hispanic black | 14 | 12 | 18 | 17 | 61
  Asian | 1 | 0 | 0 | 0 | 1
  Hispanic | 5 | 4 | 1 | 4 | 14
Insurance Coverage [Count of Participants; unit: Participants]
  Commericial | 17 | 23 | 26 | 26 | 92
  Medicare | 12 | 7 | 8 | 12 | 39
  Medicaid | 14 | 15 | 12 | 6 | 47
  Uninsured | 1 | 1 | 0 | 2 | 4
Heart Failure Classification [Count of Participants; unit: Participants] — Ejection Fraction of > or = 50% was defined as heart failure with preserved ejection fraction (HFpEF). Ejection Fraction of <50% was defined as heart failure with reduced ejection fraction (HFrEF). Where possible, this diagnosis was confirmed via physician's assessment during a patient's clinic visit within 30 days of enrollment (via medical record review by the study team).
  Participants
    (Heart failure with reduced ejection fraction HFrEF) | 36 | 33 | 30 | 29 | 128
    Heart failure with preserved ejection fraction (HFpEF) | 8 | 13 | 16 | 17 | 54
Ejection Fraction, median [Median (Inter-Quartile Range); unit: Percent of ventricular ejection] | 32 [23 to 40] | 29.5 [25 to 55] | 43.5 [29 to 52.5] | 40 [30 to 55] | 36 [26 to 49]
New York Heart Association (NYHA) classification [Count of Participants; unit: Participants] — NYHA classification is based on physician classification as described in the subject's medical record. This places patients in one of four categories based on physical limitation:
  I - No limitation of physical activity II- Slight limitation of physical activity; ordinary activity results in fatigue, palpitations, dyspnea.
  III-Marked limitation of physical activity; less than ordinary activity causes fatigue, palpitations, dyspnea.
  IV- Unable to carry on any physical activity without discomfort; symptoms of heart failure at rest.
  Participants
    Class I | 3 | 2 | 2 | 4 | 11
    Class II | 17 | 12 | 12 | 13 | 54
    Class III | 19 | 32 | 30 | 22 | 103
    Unknown | 5 | 0 | 2 | 7 | 14
Cardiac Device [Count of Participants; unit: Participants]
  Pacemaker | 5 | 7 | 6 | 1 | 19
  Implantable cardioverter defibrillator (ICD) | 11 | 16 | 15 | 19 | 61
  CardioMEMS | 1 | 2 | 2 | 4 | 9
  Other | 0 | 0 | 3 | 1 | 4
  No device | 27 | 24 | 23 | 25 | 99
Comorbidities [Count of Participants; unit: Participants]
  Diabetes Mellitus | 17 | 21 | 19 | 19 | 76
  Chronic Kidney Disease (CKD) | 6 | 12 | 9 | 11 | 38
  Chronic obstructive pulmonary disease (COPD) | 4 | 10 | 9 | 7 | 30
  Hypertension | 23 | 35 | 37 | 36 | 131
  Malignancy | 0 | 3 | 5 | 4 | 12
  Depression | 7 | 14 | 8 | 7 | 36
  Liver Disease | 0 | 0 | 0 | 1 | 1
  Coronary artery disease (CAD) | 11 | 21 | 13 | 13 | 58
  Hyperlipidemia | 18 | 17 | 21 | 12 | 68
  Obesity | 17 | 18 | 18 | 17 | 70
Medications [Count of Participants; unit: Participants]
  Beta Blocker | 41 | 40 | 41 | 42 | 164
  ACEi/ARB/ARNI | 34 | 35 | 28 | 33 | 130
  MRA | 23 | 22 | 26 | 21 | 92
  SGLT2i | 14 | 10 | 15 | 14 | 53
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1.08 [0.98 to 1.35] | 1.18 [0.93 to 1.5] | 1.15 [1.01 to 1.39] | 1.09 [0.97 to 1.35] | 1.1 [0.97 to 1.39]
Estimated Glomerular Filtration Rate (eGFR) [Median (Inter-Quartile Range); unit: mL/min/1.73m2] | 60 [55 to 60] | 59 [45 to 60] | 60 [50 to 60] | 60 [54 to 60] | 60 [50 to 60]
Potassium [Median (Inter-Quartile Range); unit: mmol/L] | 4.3 [4 to 4.6] | 4.2 [3.9 to 4.5] | 4.4 [4 to 4.6] | 4.4 [4 to 4.6] | 4.3 [4 to 4.6]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 12.7 [12 to 14.2] | 12.7 [11.4 to 14.2] | 11.9 [10.8 to 13.8] | 12.8 [11.8 to 14] | 12.7 [11.4 to 14]
White Blood Cell (WBC) Count [Median (Inter-Quartile Range); unit: 10^3 cells/µL] | 7.1 [6.2 to 9.1] | 7 [5.6 to 9] | 6.9 [6.1 to 8.1] | 7.5 [5.8 to 9.5] | 7.1 [5.8 to 8.7]
Brain Natriuretic Peptide (BNP) [Median (Inter-Quartile Range); unit: pg/mL] | 995.5 [332 to 3967] | 876.5 [490 to 2600] | 737.5 [262 to 2137.5] | 914.2 [264.5 to 2560.5] | 858 [311 to 2680]
Platelet count [Median (Inter-Quartile Range); unit: 10^3 cells/µL] | 234 [191.5 to 283] | 261.5 [205 to 323] | 218 [180 to 278] | 230 [189 to 283] | 234 [192 to 296]
Aspartate aminotransferase (AST) [Median (Inter-Quartile Range); unit: U/L] | 27 [19 to 37] | 25 [20 to 33] | 25 [19 to 32] | 28 [23 to 36] | 26 [20 to 34]
Alanine transaminase (ALT) [Median (Inter-Quartile Range); unit: U/L] | 31 [22 to 47] | 22 [15 to 33.5] | 24 [16 to 34] | 25 [19 to 38] | 25 [18 to 36]
Total Bilirubin [Median (Inter-Quartile Range); unit: Mg/dL] | 0.5 [0.4 to 0.7] | 0.3 [0.2 to 0.5] | 0.5 [0.4 to 0.7] | 0.4 [0.3 to 0.5] | 0.5 [0.3 to 0.6]
International Normalized Ratio (INR) [Median (Inter-Quartile Range); unit: Ratio] | 1.1 [1 to 1.3] | 1.1 [1 to 1.4] | 1.1 [1 to 1.2] | 1.1 [1 to 1.3] | 1.1 [1 to 1.2]
Prothrombin time (PT) [Median (Inter-Quartile Range); unit: seconds] | 11.3 [10.9 to 13.8] | 11.9 [11.1 to 14.2] | 12.1 [11.2 to 14.2] | 11.7 [11 to 12.4] | 11.9 [11.1 to 13.9]
Partial Thromboplastin Time (PTT) [Median (Inter-Quartile Range); unit: seconds] | 30.8 [26.5 to 40.2] | 25.6 [24.5 to 28.9] | 27.1 [23.9 to 44.6] | 27.5 [25.9 to 36.2] | 27.2 [25.6 to 37.3]

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life at 90 Days Post Enrollment
Description: Assessed by the change in score of the Kansas City Cardiomyopathy Questionnaire (KCCQ) survey between baseline scoring (at enrollment) and at 90 days post-enrollment. This survey is a 23 item self-administered instrument used to quantify a patient's perception of health status. For each domain reported, an overall summary scored is derived and transformed to a score range of 0-100. The Total Symptom score is the mean of the Symptom Frequency and Symptom Burden scores. The Overall Summary Score is the mean of the Physical Limitation, Total Symptom, Quality of Life and Social Limitation Scores. The Clinical Summary score is the mean of the Physical Limitation and Total Symptom scores. All KCCQ scores are summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Time Frame: Day 90 after enrollment
Measure: Median (Inter-Quartile Range); unit: Scores on a scale (difference)
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 36 | 39 | 38 | 38
Scores on a scale (difference)
  Physical Limitation | -4.2 [-14.6 to 4.2] | -4.2 [-12.5 to 4.2] | 0 [-4.2 to 10.4] | -4.2 [-16.7 to 0]
  Symptom Stability | 0 [-25 to 0] | 0 [-25 to 0] | 0 [-25 to 25] | 0 [0 to 0]
  Symptom Frequency | -2.1 [-13.5 to 10.4] | 0 [-8.3 to 10.4] | 0 [-4.2 to 18.8] | 3.1 [-4.2 to 12.5]
  Symptom Burden | 0 [-8.3 to 8.3] | 0 [-8.3 to 16.7] | 8.3 [0 to 16.7] | 0 [-8.3 to 16.7]
  Total Symptom Score | -1 [-13.5 to 7.8] | 0 [-4.2 to 14.6] | 4.2 [-1 to 16.7] | 1 [-6.2 to 12.5]
  Self-Efficacy | 0 [0 to 12.5] | 0 [0 to 12.5] | 0 [-12.5 to 12.5] | 0 [0 to 12.5]
  Quality of Life | 8.3 [-16.7 to 25] | 8.3 [-8.3 to 25] | 4.2 [-8.3 to 16.7] | 0 [-8.4 to 16.7]
  Social Limitation | 0 [-16.7 to 8.3] | 0 [-12.5 to 18.8] | 0 [-6.3 to 25] | 0 [-12.5 to 6.3]
  Clinical Summary Score | -3.1 [-10.2 to 3] | 0 [-6.2 to 7.3] | 2.8 [-1 to 14.6] | -1.6 [-10.4 to 6.3]
  Overall Summary Score | 0.3 [-9.2 to 9.4] | 2.1 [-7.8 to 14.6] | 3.4 [-2.8 to 15.1] | 2.1 [-9.1 to 6.8]

2. Secondary Outcome: Change in Quality of Life at 180 Days Post Enrollment
Description: Assessed by the change in score of the Kansas City Cardiomyopathy Questionnaire (KCCQ) survey between day 90 post enrollment and at day 180 post enrollment. This survey is a 23 item self-administered instrument used to quantify a patient's perception of health status. For each domain reported, an overall summary scored is derived and transformed to a score range of 0-100. The Total Symptom score is the mean of the Symptom Frequency and Symptom Burden scores. The Overall Summary Score is the mean of the Physical Limitation, Total Symptom, Quality of Life and Social Limitation Scores. The Clinical Summary score is the mean of the Physical Limitation and Total Symptom scores. All KCCQ scores are summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Time Frame: 180 days post enrollment
Measure: Median (Inter-Quartile Range); unit: Scores on a scale (difference)
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Scores on a scale (difference)
  Physical Limitation | -4.2 [-12.5 to 4.2] | -8.3 [-18.8 to 0] | -2.1 [-10.4 to 8.3] | -2.1 [-8.3 to 8.3]
  Symptom Stability | 0 [-25 to 0] | 0 [0 to 0] | 0 [-25 to 0] | 0 [-25 to 0]
  Symptom Frequency | 0 [-8.3 to 8.3] | 0 [-8.3 to 4.2] | 6.3 [-4.2 to 29.2] | 0 [-4.2 to 12.5]
  Symptom Burden | 0 [-8.3 to 16.7] | 0 [-16.7 to 16.7] | 0 [-8.3 to 16.7] | 0 [-16.7 to 8.3]
  Total Symptom Score | 0 [-8.3 to 10.4] | 0 [-10.4 to 6.2] | 7.3 [0 to 18.7] | 0 [-18.8 to 10.4]
  Self- Efficacy | 0 [0 to 12.5] | 0 [0 to 12.5] | 0 [0 to 12.5] | 0 [0 to 12.5]
  Quality of Life | 8.3 [0 to 16.7] | 0 [-8.3 to 8.3] | 0 [-16.7 to 16.7] | 0 [-8.3 to 25]
  Social Limitation | 0 [-9.4 to 12.5] | 0 [-12.5 to 12.5] | -3.1 [-18.8 to 5.2] | 0 [-12.5 to 16.7]
  Clinical Summary Score | -1 [-10.4 to 4.2] | -3.1 [-8.3 to 1] | 1 [-4.2 to 15.5] | -1 [-10.4 to 10.4]
  Overall Summary Score | 3.6 [-4.2 to 9.8] | 0 [-9.6 to 6.8] | -1 [-7.3 to 16.1] | 0 [-7.8 to 10.4]

3. Secondary Outcome: Number of Participants With Hospital Admission at 90 Days Post Enrollment
Description: Via medical record review. Number of patients with a hospital admission between enrollment to day 90 post enrollment.
Time Frame: 90 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants
  Participants with hospital admission | 11 | 16 | 14 | 17
  Participants with hospital admission related to congestive heart failure (CHF) | 4 | 6 | 2 | 3

4. Secondary Outcome: Number of Participants With Hospital Admission at 180 Days Post Enrollment
Description: Via medical record review. This measure is calculated as the number of participants with a hospital admission from day 90 to day 180 post enrollment.
Time Frame: 180 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants
  Participants with hospital admission | 10 | 15 | 15 | 14
  Participants with hospital admission related to CHF | 3 | 5 | 3 | 4

5. Secondary Outcome: Prescribing of Guideline-directed Medical Therapy
Description: Documented prescription or change in dosing of any one of the following medication classes: beta blockers, ACEi/ARBs, and/or spironolactone; assessed via Surescripts data collection.
Time Frame: 90 days post enrollment
Population: Surescripts data was not made available to investigators, thus we are unable to collect prescription-related data to assess this outcome.
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Prescribing of Guideline-directed Medical Therapy
Description: as for outcome 5
Time Frame: 180 days post enrollment
Population: as for outcome 5
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects Using Guideline-directed Medical Therapy at 90 Days Post Enrollment
Description: Number of patients having documented prescription of all of the following medication classes between enrollment and day 90 post enrollment: beta blockers, angiotensin-converting enzyme inhibitors (ACEi)/angiotensin receptor blockers (ARBs)/angiotensin receptor-neprilysin inhibitors (ARNI), sodium/glucose cotransporter-2 inhibitors (SGLT2i) and aldosterone receptor antagonists (MRAs); assessed via Surescripts data collection.
Time Frame: 90 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants
  Beta-blocker | 42 | 39 | 41 | 42
  ACEi/ARB/ARNI | 32 | 36 | 33 | 30
  MRA | 25 | 25 | 26 | 21
  SGLT2i | 15 | 13 | 18 | 17

8. Secondary Outcome: Number of Subjects Using Guideline-directed Medical Therapy at 180 Days Post Enrollment
Description: Number of patients having documented prescription of all of the following medication classes between day 90 post enrollment and day 180 post enrollment: beta blockers, angiotensin-converting enzyme inhibitors (ACEi)/angiotensin receptor blockers (ARBs)/angiotensin receptor-neprilysin inhibitors (ARNI), sodium/glucose cotransporter-2 inhibitors (SGLT2i) and aldosterone receptor antagonists (MRAs); assessed via Surescripts data collection.
Time Frame: 180 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants
  Beta Blocker | 40 | 38 | 40 | 40
  ACEi/ARB/ARNI | 34 | 35 | 32 | 32
  MRA | 23 | 24 | 24 | 25
  SGLT2i | 17 | 13 | 17 | 17

9. Secondary Outcome: Number of Participants With Emergency Department (ED) Visits at 90 Days Post Enrollment
Description: Via medical record review. Number of participants with an emergency department visit between enrollment and day 90 post enrollment.
Time Frame: 90 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants
  Participants with ED visit | 10 | 12 | 10 | 14
  Participants with ED visit related to CHF | 4 | 3 | 4 | 4

10. Secondary Outcome: Number of Participants With Emergency Department Visits at 180 Days Post Enrollment
Description: Via medical record review. Number of participants with an emergency department visit between day 90 and day 180 post enrollment.
Time Frame: 180 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants
  Participants with ED visit | 8 | 12 | 13 | 13
  Participants with ED visit related to CHF | 4 | 3 | 4 | 1

11. Secondary Outcome: Number of Participants With Acute Kidney Injury (AKI) Development at 90 Days Post Enrollment
Description: Via medical record review, defined as an increase in serum creatinine by 50% over baseline (pre-enrollment creatinine) at any point between enrollment day 90 post enrollment.
Time Frame: 90 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants | 4 | 6 | 2 | 6

12. Secondary Outcome: Number of Participants With Acute Kidney Injury (AKI) Development at 180 Days Post Enrollment
Description: Via medical record review, defined as an increase in serum creatinine by 50% over baseline (pre-enrollment creatinine) at any point between day 90 and day 180 post enrollment.
Time Frame: 180 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants | 3 | 2 | 3 | 3

13. Secondary Outcome: Mortality Rate at 90 Days Post Enrollment
Description: Via medical record review. Number of deaths between enrollment and 90 days post enrollment.
Time Frame: 90 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants | 0 | 0 | 0 | 1

14. Secondary Outcome: Mortality Rates at 180 Days Post Enrollment
Description: Via medical record review. Number of deaths between day 90 and day 180 post enrollment.
Time Frame: 180 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants | 1 | 2 | 0 | 1

15. Secondary Outcome: Number of Participants With at Least One Clinic No-show at 90 Days Post Enrollment
Description: Via medical record review; number of participants with at least one clinic no show between enrollment and day 90 post enrollment.
Time Frame: 90 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants | 12 | 12 | 8 | 10

16. Secondary Outcome: Number of In-person and Remote Clinic Visits at 90 Days Post Enrollment
Description: Via medical record review. Number of visits between enrollment and 90 days post enrollment.
Time Frame: 90 days post enrollment
Measure: Median (Inter-Quartile Range); unit: Clinic visits
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Clinic visits
  Number of in-person clinic visits | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
  Number of virtual/phone clinic visits | 1 [1 to 1] | 1 [1 to 2] | 2 [1 to 4] | 1 [1 to 2]

17. Secondary Outcome: Number of In-person and Remote Clinic Visits at 180 Days Post Enrollment
Description: Via medical record review. Number of visits between day 90 and day 180 post enrollment.
Time Frame: 180 days post enrollment
Measure: Median (Inter-Quartile Range); unit: Clinic visits
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Clinic visits
  Number of in-person clinic visits | 1 [0 to 1] | 0 [0 to 1] | 1 [0 to 2] | 0 [0 to 1]
  Number of virtual/phone clinic visits | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

18. Secondary Outcome: Number of Remote Device Checks by Providers at 90 Days Post Enrollment
Description: Via medical record review
Time Frame: 90 days post enrollment
Measure: Median (Inter-Quartile Range); unit: Remote device checks
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Remote device checks | 17 [5 to 29] | 1 [1 to 3] | 3 [3 to 3] | 6 [5 to 8]

19. Secondary Outcome: Number of Remote Device Checks by Providers at 180 Days Post Enrollment
Description: Via medical record review
Time Frame: 180 days post enrollment
Measure: Median (Inter-Quartile Range); unit: Remote device checks
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Remote device checks | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

20. Secondary Outcome: Number of Phone Calls Between Provider and Participant at 90 Days Post Enrollment
Description: Via medical record review of telephone logs between enrollment and day 90 post enrollment.
Time Frame: 90 days post enrollment
Measure: Median (Inter-Quartile Range); unit: Provider-Participant calls
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Provider-Participant calls
  Number of calls to clinic with questions/inquiry for provider | 1 [1 to 4] | 1 [1 to 2] | 1 [1 to 2] | 2 [1 to 3]
  Number of calls by provider/clinic to patient for check-in | 2 [1 to 4] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 5]
  Number of calls by provider/clinic to patient with test results | 2 [1 to 2] | 2 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
  Number of appointment reminder calls made to patient | 3 [1 to 4] | 2 [1 to 3] | 2 [1 to 2] | 2 [1 to 2]

21. Secondary Outcome: Number of Phone Calls Between Provider and Participant at 180 Days Post Enrollment
Description: Via medical record review of telephone logs
Time Frame: 180 days post enrollment
Measure: Median (Inter-Quartile Range); unit: Patient-provider calls
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Patient-provider calls
  Number of calls to clinic with questions/inquiry for provider | 0 [0 to 0] | 0 [0 to 1] | 0 [0 to 0] | 0 [0 to 1]
  Number of calls by provider/clinic to patient for check-in | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]
  Number of calls by provider/clinic to patient with test results | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Number of appointment reminder calls made to patient | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]

22. Secondary Outcome: Average Time Devoted by Provider to Patient Care
Description: Via medical record review of chart openings per patient
Time Frame: 90 days post enrollment
Population: Current EHR infrastructure does not capture chart openings, thus outcome cannot be assessed because data not collected.
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Average Time Devoted by Provider to Patient Care
Description: Via medical record review of chart openings per patient
Time Frame: 180 days post enrollment
Population: Current EHR infrastructure does not capture chart openings, thus outcome cannot be assessed because data not collected.
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects Who Complete on Boarding and Baseline Assessments
Description: Collected from patient enrollment platform
Time Frame: Within one week of consent
Measure: Count of Participants; unit: Participants
Arm/Group | Control | BodyPort | Noom | Conversa
Number analyzed (Participants) | 44 | 46 | 46 | 46
Participants | 44 | 46 | 46 | 46

25. Secondary Outcome: Number of Subjects Who Complete Digital Health Product Set up
Description: Assessed as number of subjects who used device at least once during their duration in the study, up to 90 days post enrollment.
Time Frame: 90 days post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | BodyPort | Noom | Conversa
Number analyzed (Participants) | 46 | 46 | 46
Participants | 43 | 23 | 33

26. Secondary Outcome: Number of Weekly Interactions With the Device
Description: Information collected from device metrics to assess frequency of use
Time Frame: 90 days post enrollment
Measure: Mean (Standard Deviation); unit: Weekly interactions with device
Arm/Group | BodyPort | Noom | Conversa
Number analyzed (Participants) | 46 | 46 | 46
Weekly interactions with device
  Week 1 | 4 (2.2) | 6.9 (5.5) | 1.8 (0.5)
  Week 2 | 8.1 (5.9) | 6.1 (1.8) | 1 (.2)
  Week 3 | 7.7 (5.4) | 5.7 (2.2) | 1 (0)
  Week 4 | 8.3 (7.5) | 5.9 (2.1) | 1 (.2)
  Week 5 | 6.8 (3.7) | 5.7 (2.2) | 1 (.2)
  Week 6 | 6.5 (3) | 6.6 (1.4) | 1 (.2)
  Week 7 | 6.5 (2.7) | 6 (1.9) | 1 (0.2)
  Week 8 | 6.3 (3.1) | 6.8 (.6) | 1.1 (.3)
  Week 9 | 5.7 (3.3) | 5.4 (2.5) | 1 (.2)
  Week 10 | 5.9 (3.6) | 5.5 (2.5) | 1 (.2)
  Week 11 | 6.3 (2.8) | 6.4 (1.9) | 1.1 (0.3)
  Week 12 | 6.3 (3.2) | 5.8 (2.4) | 1 (0)

27. Secondary Outcome: Number of Weekly Interactions With the Device
Description: Information collected from device metrics to assess frequency of use
Time Frame: 180 days post enrollment
Measure: Mean (Standard Deviation); unit: Weekly interactions with device
Arm/Group | BodyPort | Noom | Conversa
Number analyzed (Participants) | 46 | 46 | 46
Weekly interactions with device
  Week 13 | 6 (3.2) | 6.5 (1.5) | 1 (.2)
  Week 14 | 6.9 (3.6) | 5.8 (2.2) | 1 (.2)
  Week 15 | 6.3 (2.3) | 6.6 (1.3) | 1 (0)
  Week 16 | 5.5 (2.7) | 6.7 (.9) | 1.2 (.5)
  Week 17 | 6.1 (2.9) | 5.8 (2.1) | 1.1 (.3)
  Week 18 | 5.6 (2.8) | 6.8 (.4) | 1.1 (.3)
  Week 19 | 5.9 (3.3) | 6.5 (1.8) | 1 (.2)
  Week 20 | 6.3 (2.8) | 6.8 (.7) | 1 (.2)
  Week 21 | 5.2 (2.5) | 6.4 (1.3) | 1.1 (.3)
  Week 22 | 5.5 (2.6) | 6.4 (1.8) | 1.2 (.4)
  Week 23 | 5.2 (3.3) | 6.3 (1.6) | 1 (.2)
  Week 24 | 5.2 (3.3) | 6.3 (1.6) | 1 (.2)

28. Secondary Outcome: Average Number of Daily Interactions With the Device
Description: Information collected from device metric to assess frequency of use
Time Frame: 90 days post enrollment
Measure: Mean (Standard Deviation); unit: Interactions per day with device
Arm/Group | BodyPort | Noom | Conversa
Number analyzed (Participants) | 46 | 46 | 46
Interactions per day with device | .7 (.4) | .5 (.4) | .1 (.04)

29. Secondary Outcome: Average Number of Daily Interactions With the Device
Description: Information collected from device metric to assess frequency of use
Time Frame: 180 days post enrollment
Measure: Mean (Standard Deviation); unit: Daily interactions with device
Arm/Group | BodyPort | Noom | Conversa
Number analyzed (Participants) | 46 | 46 | 46
Daily interactions with device | .6 (.4) | .9 (.8) | .2 (.09)

ADVERSE EVENTS:
Time Frame: Duration of a subject's participation, up to 180 days post enrollment.
Arm/Group | Control | BodyPort | Noom | Conversa
All-Cause Mortality (participants affected / at risk) | 1/44 | 2/46 | 0/46 | 2/46
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/44 | 0/46 | 0/46 | 0/46

LIMITATIONS AND CAVEATS:
* Exclusion of patients over 80 years of age, which could intrinsically bias the trial towards those with more digital literacy.
* A proportion of participants randomized to each of the groups that decided not to use the technology during their follow-up period. Our intention to treat analysis sought to evaluate real-world use and applicability.
* The study was conducted across eleven outpatient HF clinics within a large health system in CT, USA, which could limit generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT04394754/Prot_SAP_000.pdf